CLINICAL TRIAL: NCT01856829
Title: Effect of Omega-3 Phospholipids on Attentional Abilities and Perceptual-cognitive Training
Brief Title: Effect of Omega-3 Phospholipids on Perceptual-cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Neptune Technologies and Bioressources Inc. (Industry)
Responsible Party: Principal Investigator, Jocelyn Faubert, Full Professeur, Université de Montréal
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: NKO-PC_01
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Cognition - Other
MeSH Terms: interventions — Docosahexaenoic Acids; Plant Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control participants will take placebo capsules daily for 4 weeks before and for the duration of the test. At week 4, participants will undergo a training protocol consists of a series of five sessions consecutively performed at intervals of 3 to 7 days. Taking products will be made more specifically 30 minutes before the start of the sessions.
  Interventions: Other: Placebo
- Omega-3 (Experimental): Omega-3 participants will take capsules daily for 4 weeks before and for the duration of the test. At week 4, participants will undergo a training protocol consists of a series of five sessions consecutively performed at intervals of 3 to 7 days. Taking products will be made more specifically 30 minutes before the start of the sessions.
  Interventions: Dietary Supplement: Omega-3

INTERVENTIONS:
Dietary Supplement: Omega-3 — The capsule will be take daily for 4 weeks before and for the duration of the tests of the perceptual-cognitive training protocol. The testing period will held at intervals of 3 to 7 days for 5 sessions (maximum of 5 weeks testing). Taking products will be made more specifically 30 minutes before the start of the sessions.
  Other Names: health Canada product number 80006416
  Arms: Omega-3
Other: Placebo — The capsule will be take daily for 4 weeks before and for the duration of the tests of the perceptual-cognitive training protocol. The testing period will held at intervals of 3 to 7 days for 5 sessions (maximum of 5 weeks testing). Taking products will be made more specifically 30 minutes before the start of the sessions.
  Other Names: vegetable oil
  Arms: Control

SUMMARY:
Omega 3 in the form of phospholipids are the main component of nerve cells and their oral intake is known to have a positive impact on behavior disorders such as depression or bipolar disorder. Their consumption would improve brain function while increasing the ability to concentrate. The study aims to determine the effect of an increase in Omega 3 in the form of phospholipids on the processing of visual information in the brain and in particular the attention and perceptual-cognitive learning in a three dimensions environment. Eighty subjects (40 young (18-35 years) and 40 older (60-75 years)) divided into four groups, two Omega-3 (20 young and 20 older) and two other placebo (20 young and 20 elderly ), will in this study, performing a complex perceptual-cognitive task such as the pursuit of moving objects in a 3D space. This stimulus was chosen because it is very similar to the situations of daily life, but also because it involves a mechanism of perceptual-cognitive level. The main objective is to demonstrate the positive effect of Omega-3 phospholipids on the perceptual-cognitive training.

DETAILED DESCRIPTION:
Improve visual skills through training and perceptual-cognitive learning could be a method aimed to repair partial neurophysiological deficits or produce new brain networks. Studies suggest that the mechanisms of attention and cortical plasticity have a role to play in information retrieval. In addition, he has been shown that Omega 3 in the form of phospholipids are the main component of nerve cells and taken orally makes a positive impact on behavior disorders such as depression or bipolar disorder. Their consumption would also help improve brain function while increasing the ability to concentrate.

The perceptual-cognitive ability is a very high level treatment of complex visual information. However, this ability only has our brain seems to be driven by the fact that the brain has great plasticity. This means that there is a neuronal reorganization in learning new capacity. 3D-MOT, or 3-Dimensional Multiple Object Tracking is a technique that allows the study of the visual system for tracking moving targets in 3D. It is a task of multifocal attentional pursuit which assesses the ability to keep the position of different moving targets from other similar objects. Performance is measured based on the number of objects that have been successfully followed. Previous studies have also shown that most young patients can typically take four objects simultaneously. In addition, this tracking capability, when speed is used as the dependent variable seems drivable. Therefore, Faubert and Sidebottom have shown that young people could significantly increase their speed thresholds. Legault and Faubert (2012) have demonstrated that training with the method of 3D-MOT generates significant improvements in visual-cognitive abilities as the perception of movement of the human body, a crucial index to avoid collisions when we navigate in a dense crowd for example.

The purpose of this project is to evaluate the impact of taking Omega-3 phospholipid form on perceptual-cognitive abilities, on the learning rate (curve) of young and older adults. The sample is composed of 40 young people (20 to 35) and 40 older adults (60-75) divided into two groups. The stimulus will be a task of multiple objects or 3D-MOT that consist to simultaneously track multiple moving objects among distractors, all will be presented on a 3D television screen . The performance of the observer (speed thresholds) will be evaluated based on three elements followed without error.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 or from 60 to 75 years;
* binocular visual acuity greater or equal to 6/6 (Snellen), with or without correction;
* Stereoacuity greater than 40 second of arc measured by the Frisby Stereo acuity test; Visual Field without anomalies or constriction;
* Scores for the mini-mental-state-examination(elderly person only) greater than 24/30
* Good general health

Exclusion Criteria:

* If you are taking medication acting on vigilance and attention;
* If you suffer from any eye diseases (glaucoma, age-related macular degeneration, diabetic retinopathy);
* If you suffer from postural balance disorders.
* If you suffer from chronic or severe diseases, including neurological disorders (eg epilepsy).
* If you are an elite athlete.
* If you eat fish or seafood more than 2 times per week;
* If you play at video games 3 hours or more per day / 5 days a week or more.
* If you suffer from allergy to fish or seafood
* If you consumed or have consumed in the previous 3 months, food supplements based on omega-3 (eg oil of fish or Krill Oil)
* If you have a blood coagulation disorder, or are receiving anticoagulant therapy.
* If you have participated in a clinical study in a period shorter than four weeks
* If you do not understand the constraints of the study.
* If you refuse to give your written consent.
* If you are pregnant or breastfeeding.
* If you got a speed threshold 40% higher than the group average, in the first session tracking targets.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Speed-thresholds performance | 6 weeks
  We will measure speed thresholds performance on a perceptual-cognitive task while participants will take Omega-3 or a placebo. Products comply with applicable regulations by Health Canada (80033441). The participants will take capsule daily for 4 weeks before and for the duration of the perceptual-cognitive training protocol. Participant will not be inform on the nature of their capsule (Omega-3 or placebo). All participants will undergo a training protocol that consists of a series of five sessions performed at intervals of 3 to 7 days. The product will be taken 30 minutes before the start of the sessions. During the sessions, participants will perform a 3D-multiple object tracking task. The stimulus consists to simultaneously track multiple moving objects among distractors and we measured the maximum speed at which the objects could travel, for younger and older observers to complete the task with no errors.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Faubert, PhD, Study Chair — École d'optométrie, Université de Montréal
Locations (2):
- Canada (2):
  - Visual psychophysics and perception laboratory, Montreal, Quebec
  - École d'optométrie, Université de Montréal, Montreal, Quebec

REFERENCES:
- [Background] Alvarez GA, Franconeri SL. How many objects can you track? Evidence for a resource-limited attentive tracking mechanism. J Vis. 2007 Oct 30;7(13):14.1-10. doi: 10.1167/7.13.14. PMID 17997642
- [Background] Bloch MH, Qawasmi A. Omega-3 fatty acid supplementation for the treatment of children with attention-deficit/hyperactivity disorder symptomatology: systematic review and meta-analysis. J Am Acad Child Adolesc Psychiatry. 2011 Oct;50(10):991-1000. doi: 10.1016/j.jaac.2011.06.008. Epub 2011 Aug 12. PMID 21961774
- [Background] Draganski B, May A. Training-induced structural changes in the adult human brain. Behav Brain Res. 2008 Sep 1;192(1):137-42. doi: 10.1016/j.bbr.2008.02.015. Epub 2008 Feb 17. PMID 18378330
- [Background] Legault I, Faubert J. Perceptual-cognitive training improves biological motion perception: evidence for transferability of training in healthy aging. Neuroreport. 2012 May 30;23(8):469-73. doi: 10.1097/WNR.0b013e328353e48a. PMID 22495038
- [Background] Pylyshyn Z. The role of location indexes in spatial perception: a sketch of the FINST spatial-index model. Cognition. 1989 Jun;32(1):65-97. doi: 10.1016/0010-0277(89)90014-0. PMID 2752706
- [Background] Sabel BA, Henrich-Noack P, Fedorov A, Gall C. Vision restoration after brain and retina damage: the "residual vision activation theory". Prog Brain Res. 2011;192:199-262. doi: 10.1016/B978-0-444-53355-5.00013-0. PMID 21763527
- [Background] Sarris J, Mischoulon D, Schweitzer I. Omega-3 for bipolar disorder: meta-analyses of use in mania and bipolar depression. J Clin Psychiatry. 2012 Jan;73(1):81-6. doi: 10.4088/JCP.10r06710. Epub 2011 Aug 9. PMID 21903025
- [Background] Sublette ME, Ellis SP, Geant AL, Mann JJ. Meta-analysis of the effects of eicosapentaenoic acid (EPA) in clinical trials in depression. J Clin Psychiatry. 2011 Dec;72(12):1577-84. doi: 10.4088/JCP.10m06634. Epub 2011 Sep 6. PMID 21939614
- [Background] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038
- [Background] Faubert J, Sidebottom L. Perceptual-cognitive training of athletes. Journal of clinical sports psychology (6):85-102, 2012.